CLINICAL TRIAL: NCT04982588
Title: Medtronic CoreValve™ Evolut™ PRO System China Clinical Study
Brief Title: Evolut PRO China Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT18065EVR009
Record Dates: First submitted 2021-07-08; First posted 2021-07-29 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Severe, Symptomatic Aortic Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medtronic CoreValve™ Evolut™ PRO System (Experimental): The system comprised of the following three components:
  1. CoreValve™ Evolut™ PRO Transcatheter Aortic Valve (TAV)
  2. EnVeo™ PRO Delivery Catheter System (DCS)
  3. EnVeo™ PRO Loading System (LS)
  Interventions: Device: Medtronic CoreValve™ Evolut™ PRO System

INTERVENTIONS:
Device: Medtronic CoreValve™ Evolut™ PRO System — The system comprised of the following three components:
  1. CoreValve™ Evolut™ PRO Transcatheter Aortic Valve (TAV)
  2. EnVeo™ PRO Delivery Catheter System (DCS)
  3. EnVeo™ PRO Loading System (LS)

SUMMARY:
Interventional study to evaluate the safety and efficacy of the Medtronic CoreValve™ Evolut™ PRO System when used by China implanting centers in Chinese patients with severe symptomatic aortic stenosis (AS) who are at high risk for Surgical Aortic Valve Replacement (SAVR).

DETAILED DESCRIPTION:
The study is targeting 6 centers with a maximum of 8 centers in China and estimating 65 subjects with a maximum of up to 70 subjects with attempted implants including 50 subjects with an attempted implant in primary study population and the first two attempted subjects at each site for roll-in population. The subjects will follow the assessment with pre and post-procedure, discharge, 30 days(primary endpoint), 6 months, 1 year, and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aortic valve area (AVA) < 1.0 cm2 (or indexed AVA <0.6 cm2/m2) OR mean gradient > 40 mmHg, OR max aortic velocity > 4.0 m/sec
2. High risk for SAVR defined as STS-PROM score ≥ 8% AND ≤ 15%, OR documented Heart Team agreement of high risk for AVR due to frailty or comorbidities
3. Symptoms of aortic stenosis and NYHA ≥ II

Exclusion Criteria:

1. Age is less than 65 years old
2. Non-calcified aortic valve
3. Bicuspid aortic valve with no raphe or 2 raphes (Sievers classification type 0 or type 2)
4. Ascending aortic diameter > 4.5 cm

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2028-05-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Chinese PLA Medical School, Beijing, Beijing Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Medtronic CoreValve™ Evolut™ PRO System: Subjects treated with the Medtronic CoreValve™ Evolut™ PRO System.
  Primary Study Population: 52 enrolled subjects, 50 attempted implants
  The Primary Study Population Attempted Implant set (N=50)was the basis for the primary safety endpoint of the study, and the Primary Study Population Implanted set (N=49) was the basis for the assessment of the primary efficacy endpoint of the study.
Period: Overall Study
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Started | 52 (Enrolled, enrollment is defined as the Date of Eligibility Review Committee (ERC) approval)
Exited Prior to Procedure | 2
Implanted (Subjects who are implanted with the Evolut PRO) | 49
Attempted, Not Implanted | 1
Completed | 50 (Attempted, includes all subjects who are brought into the procedure room and any of the following have occurred: anesthesia administered, vascular line placed, TEE placed, or any monitoring line placed.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Primary Study Population consisted of 50 participants with an attempted implant
Groups:
- Experimental: Medtronic CoreValve™ Evolut™ PRO System: Subjects treated with the Medtronic CoreValve™ Evolut™ PRO System.
  Primary Study Population: 50 attempted implants
  The Primary Study Population Attempted Implant set (N=50)was the basis for the primary safety endpoint of the study, and the Primary Study Population Implanted set (N=49) was the basis for the assessment of the primary efficacy endpoint of the study.
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 50
BSA [Mean (Standard Deviation); unit: m^2] | 1.6 (0.2)
NYHA [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
  Participants
    I | 0
    II | 6
    III | 26
    IV | 18
STS Score [Mean (Standard Deviation); unit: %] — The Society of Thoracic Surgeons (STS) Score is a score that represents the risk of operative mortality, major morbidity, and complications for adult cardiac surgeries.
  A total STS Score, presented as a risk probability on a scale of 0-100%, is calculated based on patient characteristics.
  The STS Score is calculated before a patient undergoes the transcatheter aortic valve replacement (TAVR) index procedure in the study, and a higher STS Score means a patient is at higher risk for surgery.
  % | 5.6 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: All-cause mortality at 30 days
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0.0

2. Primary Outcome: Percentage (%) of Subjects With Evaluable Echocardiograms With Moderate or Severe Aortic Regurgitation by Transthoracic Echocardiography (TTE)
Description: Percentage (%) of Subjects with evaluable echocardiograms with moderate or severe aortic regurgitation by transthoracic echocardiography (TTE)
Time Frame: 30 days
Population: Number of subjects with evaluable aortic regurgitation from echo core lab
Measure: Number (95% Confidence Interval); unit: Percentage (%) of participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 45
Percentage (%) of participants | 2.2 [0.1 to 11.8]

3. Secondary Outcome: Incidence of an VARC II Combined Composite
Description: Incidence of an VARC II combined composite includes the following components:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury: stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number (95% Confidence Interval); unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 4 [1.0 to 15.2]

4. Secondary Outcome: Event Rates of the Individual Components of the VARC II Composite
Description: Event rate of the individual components listed in the outcome
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate)
  All-Cause Mortality | 0.0
  All Stroke | 0.0
  Life Threatening or Disabling Bleeding | 0.0
  Acute Kidney Injury: Stage 2 or 3 | 0.0
  Coronary Artery Obstruction | 4.0
  Major Vascular Complication | 0.0
  Valve-Related Dysfunction Requiring Repeat Procedure | 0.0

5. Secondary Outcome: New Permanent Pacemaker Rate
Description: New permanent pacemaker rate
Time Frame: 30 days
Population: Number of attempted implant population. Subjects with a pacemaker or ICD at baseline are excluded.
Measure: Number (95% Confidence Interval); unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 46
Percent of Participants (K-M Rate) | 8.8 [3.4 to 21.9]

6. Secondary Outcome: Device Success Rate
Description: Device success rate:
  * Percentage of participants with absence of procedural mortality, AND
  * Percentage of participants with correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
  * Percentage of participants with intended performance of the prosthetic heart valve, defined as the absence of patient-prosthesis-mismatch and mean aortic valve gradient less than 20 mmHg (or peak velocity <3m/sec), AND absence of moderate or severe prosthetic valve regurgitation
Time Frame: Between 24 hours and 7 days post procedure
Population: Number of attempted implant subjects with evaluable data for device success
Measure: Number (95% Confidence Interval); unit: Percentage (%) of participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 36
Percentage (%) of participants | 63.9 [46.2 to 79.2]

7. Secondary Outcome: Valve Performance Parameter - Mean Aortic Gradient
Description: Mean aortic gradient
Time Frame: 30 days
Population: Number of implanted subjects with echo core lab evaluable values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 43
mmHg | 10.7 (4.9)

8. Secondary Outcome: Valve Performance Parameter - Effective Orifice Area
Description: Effective orifice area
Time Frame: 30 days
Population: Number of implanted subjects with echo core lab evaluable values
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 32
cm^2 | 1.8 (0.4)

9. Secondary Outcome: Valve Performance Parameter -Degree of Aortic Regurgitation (Transvalvular, Paravalvular, Total)
Description: Degree of aortic regurgitation (transvalvular, paravalvular, total)
Time Frame: 30 days
Population: Number of implanted subjects with echo core lab evaluable values
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 45
Participants
  Total Aortic Regurgitation: None | 18
  Total Aortic Regurgitation: Trace | 15
  Total Aortic Regurgitation: Mild | 9
  Total Aortic Regurgitation: Mild to Moderate | 2
  Total Aortic Regurgitation: Moderate | 1
  Total Aortic Regurgitation: Moderate to Severe | 0
  Total Aortic Regurgitation: Severe | 0
  Paravalvular Aortic Regurgitation: None | 19
  Paravalvular Aortic Regurgitation: Trace | 14
  Paravalvular Aortic Regurgitation: Mild | 9
  Paravalvular Aortic Regurgitation: Mild to Moderate | 2
  Paravalvular Aortic Regurgitation: Moderate | 1
  Paravalvular Aortic Regurgitation: Moderate to Severe | 0
  Paravalvular Aortic Regurgitation: Severe | 0
  Transvalvular Aortic Regurgitation: None | 43
  Transvalvular Aortic Regurgitation: Trace | 2
  Transvalvular Aortic Regurgitation: Mild | 0
  Transvalvular Aortic Regurgitation: Mild to Moderate | 0
  Transvalvular Aortic Regurgitation: Moderate | 0
  Transvalvular Aortic Regurgitation: Moderate to Severe | 0
  Transvalvular Aortic Regurgitation: Severe | 0

10. Other Pre Specified Outcome: Event Rates of TAVI-related Complications
Description: Rate of the following TAVI-related complications:
  1. change to surgery
  2. need for cardiopulmonary mechanical assistance
  3. coronary occlusion or obstruction
  4. annular rupture or dissection
  5. ventricular perforation
  6. mitral valve damage
  7. prosthetic valve displacement, migration, or embolism
  8. acute kidney injury (up to 7 days post procedure)
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate)
  change to surgery | 0
  need for cardiopulmonary mechanical assistance | 0
  coronary occlusion or obstruction | 4.0
  annular rupture or dissection | 0
  ventricular perforation | 0
  mitral valve damage | 0
  prosthetic valve displacement, migration, or embolism | 2.0
  acute kidney injury | 0

11. Other Pre Specified Outcome: All-cause Mortality
Description: Percentage of participants with all-cause mortality
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 2.0

12. Other Pre Specified Outcome: All-cause Mortality
Description: Percentage of participants with all-cause mortality
Time Frame: 1 year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 8.2

13. Other Pre Specified Outcome: All Stroke
Description: Incidence of stroke (disabling and non-disabling)
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 2.0

14. Other Pre Specified Outcome: All Stroke
Description: Incidence of stroke (disabling and non-disabling)
Time Frame: 1 year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Groups:
- Experimental: Medtronic CoreValve™ Evolut™ PRO System - 1 Year: Subjects treated with the Medtronic CoreValve™ Evolut™ PRO System.
  Primary Study Population: 50 attempted implants
  The Primary Study Population Attempted Implant set (N=50)was the basis for the primary safety endpoint of the study, and the Primary Study Population Implanted set (N=49) was the basis for the assessment of the primary efficacy endpoint of the study.
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System - 1 Year
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 4.1

15. Other Pre Specified Outcome: Myocardial Infarction
Description: Incidence of MI
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 2.0

16. Other Pre Specified Outcome: Myocardial Infarction
Description: Incidence of MI
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 2.0

17. Other Pre Specified Outcome: Myocardial Infarction
Description: Incidence of MI
Time Frame: 1 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 4.1

18. Other Pre Specified Outcome: Incidence of Life-threatening Bleeding
Description: Incidence of life-threatening bleeding:
  1. Fatal bleeding (BARC type 5) OR
  2. Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC type 3b and 3c) OR
  3. Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b) OR
  4. Overt source of bleeding with drop in hemoglobin ≥5 g/dL or whole blood or packed red blood cells (RBCs) transfusion ≥4 units* (BARC type 3b)
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

19. Other Pre Specified Outcome: Incidence of Life-threatening Bleeding
Description: as for outcome 18
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

20. Other Pre Specified Outcome: Incidence of Life-threatening Bleeding
Description: as for outcome 18
Time Frame: 1 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

21. Other Pre Specified Outcome: New AV-Conduction Disturbances (Left Bundle Branch Block (LBBB) and Right Bundle Branch Block (RBBB))
Description: Incidence of either LBBB or RBBB
Time Frame: 30 days
Population: Number of attempted implant population. Subjects with LBBB or RBBB at baseline are excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 42
Participants | 5

22. Other Pre Specified Outcome: Incidence of Prosthetic Valve Endocarditis
Description: Incidence of prosthetic valve endocarditis:
  Any one of the following:
  1. Fulfillment of the following Duke criteria for definite endocarditis
     * Histologic and/or microbiologic evidence of infection at surgery or autopsy, or
     * 2 major criteria, or
     * 1 major criteria and 3 minor criteria, or
     * 5 minor criteria
  2. Evidence of abscess, paravalvular leak, pus, or vegetation confirmed as secondary to infection by histological or bacteriological studies during a re-operation
  3. Findings of abscess, pus, or vegetation involving the CoreValve™ Evolut™ PRO at autopsy
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

23. Other Pre Specified Outcome: Incidence of Prosthetic Valve Endocarditis
Description: as for outcome 22
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

24. Other Pre Specified Outcome: Incidence of Prosthetic Valve Endocarditis
Description: as for outcome 22
Time Frame: 1 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

25. Other Pre Specified Outcome: Incidence of Prosthetic Valve Thrombosis
Description: Incidence of Prosthetic valve thrombosis:
  Any thrombus attached to or near an implanted valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment.
  *Valve-associated thrombus identified at autopsy in a patient whose cause of death was not valve related should not be reported as valve thrombosis.
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

26. Other Pre Specified Outcome: Incidence of Prosthetic Valve Thrombosis
Description: as for outcome 25
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

27. Other Pre Specified Outcome: Incidence of Prosthetic Valve Thrombosis
Description: as for outcome 25
Time Frame: 1 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

28. Other Pre Specified Outcome: Valve-related Dysfunction
Description: Incidence of valve-related dysfunction defined as moderate or severe prosthetic valve stenosis, or moderate or severe prosthetic regurgitation (per VARC II)
Time Frame: 1 Year
Population: Number of implanted subjects with evaluable site-reported echo data
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 32
Participants | 1

29. Other Pre Specified Outcome: Incidence of Valve-related Dysfunction Requiring Repeat Procedure
Description: Incidence of Valve-related dysfunction requiring repeat procedure
Time Frame: 30 days
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

30. Other Pre Specified Outcome: Incidence of Valve-related Dysfunction Requiring Repeat Procedure
Description: Incidence of Valve-related dysfunction requiring repeat procedure
Time Frame: 6 months
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

31. Other Pre Specified Outcome: Incidence of Valve-related Dysfunction Requiring Repeat Procedure
Description: Incidence of Valve-related dysfunction requiring repeat procedure
Time Frame: 1 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0

32. Other Pre Specified Outcome: Valve Hemodynamic Performance Metric - Mean Aortic Gradient
Description: Mean aortic gradient
Time Frame: 1 year
Population: Number of implanted subjects with site reported echo evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 34
mmHg | 10.1 (4.5)

33. Other Pre Specified Outcome: Valve Hemodynamic Performance Metric - Effective Orifice Area
Description: Effective orifice area
Time Frame: 1 year
Population: Number of implanted subjects with site reported echo evaluable data
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 32
cm^2 | 1.68 (0.52)

34. Other Pre Specified Outcome: Valve Hemodynamic Performance Metric - Degree of Aortic Regurgitation (Transvalvular, Paravalvular, Total)
Description: Degree of aortic regurgitation (transvalvular, paravalvular, total)
Time Frame: 1 year
Population: Number of implanted subjects with site reported echo evaluable data
Measure: Count of Participants; unit: Participants
Groups:
- Total Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System; Paravalvular Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System; Transvalvular Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System: Subjects treated with the Medtronic CoreValve™ Evolut™ PRO System.
  Primary Study Population: 50 attempted implants
  The Primary Study Population Attempted Implant set (N=50)was the basis for the primary safety endpoint of the study, and the Primary Study Population Implanted set (N=49) was the basis for the assessment of the primary efficacy endpoint of the study.
Arm/Group | Total Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System | Paravalvular Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System | Transvalvular Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 34 | 34 | 34
Participants
  None | 17 | 18 | 32
  Trace | 8 | 7 | 1
  Mild | 8 | 8 | 1
  Mild to Moderate | 0 | 0 | 0
  Moderate | 1 | 1 | 0
  Moderate to Severe | 0 | 0 | 0
  Severe | 0 | 0 | 0

35. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Classification
Description: New York Heart Association (NYHA) functional classification system is a tool that classifies patients with heart failure into one of four classes according to their degree of systems at rest and with activity. Below are the four classes and the associated patient symptoms (i.e., Class I has no limitations of physical activity vs. Class IV is most symptomatic and patient has symptoms of heart failure at rest).
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: 30 days
Population: Number of attempted subjects with available NYHA
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 46
Participants
  NYHA I | 13
  NYHA II | 27
  NYHA III | 5
  NYHA IV | 1
  Died prior to visit | 0

36. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Classification
Description: as for outcome 35
Time Frame: 6 month
Population: Number of attempted subjects with available NYHA
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 47
Participants
  NYHA I | 27
  NYHA II | 17
  NYHA III | 2
  NYHA IV | 0
  Died prior to visit | 1

37. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Classification
Description: as for outcome 35
Time Frame: 1 Year
Population: Number of attempted subjects with available NYHA
Measure: Count of Participants; unit: Participants
Groups:
- Medtronic CoreValve™ Evolut™ PRO System: Subjects treated with the Medtronic CoreValve™ Evolut™ PRO System. Primary Study Population: 50 attempted implants The Primary Study Population Attempted Implant set (N=50)was the basis for the primary safety endpoint of the study, and the Primary Study Population Implanted set (N=49) was the basis for the assessment of the primary efficacy endpoint of the study.
Arm/Group | Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 39
Participants
  NYHA I | 12
  NYHA II | 19
  NYHA III | 4
  NYHA IV | 0
  Died Prior to visit | 4

38. Other Pre Specified Outcome: EQ-5D Quality of Life
Description: EuroQol Group developed this Quality of Life (QOL) questionnaire referred to as EQ-5D that includes a descriptive system comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
  The answers given to ED-5D can be converted into EQ-5D index and utility scores anchored at 0 for death and 1 for perfect health.
  The EQ-5D Index Score is calculated for each study participant and the descriptive statistical summary of the EQ-5D score for the study population is provided.
  The EQ-5D Visual Analog Scale (VAS) Score is a scale numbered 0 to 100 (0 is the worse health the patient can imagine and 100 is the best health the patient can imagine).
Time Frame: 30 days
Population: Number of attempted subjects with available EQ5D
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 46
Score on a scale
  EQ-5D Index Score | 0.880 (0.095)
  EQ-5D VAS Score | 79.1 (14.7)

39. Other Pre Specified Outcome: EQ-5D Quality of Life
Description: as for outcome 38
Time Frame: 1 Year
Population: Number of attempted subjects with available EQ5D
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 34
Score on a scale
  EQ-5D Index Score | 0.905 (0.093)
  EQ-5D VAS Score | 79.8 (10.4)

40. Other Pre Specified Outcome: All-cause Mortality
Description: Percentage of participants with all-cause mortality
Time Frame: 2 year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 10.3

41. Other Pre Specified Outcome: All Stroke
Description: Incidence of stroke (disabling and non-disabling)
Time Frame: 2 year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System - 1 Year
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 6.4

42. Other Pre Specified Outcome: Myocardial Infarction
Description: Incidence of MI
Time Frame: 2 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 4.1

43. Other Pre Specified Outcome: Incidence of Life-threatening Bleeding
Description: as for outcome 18
Time Frame: 2 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0.0

44. Other Pre Specified Outcome: Incidence of Prosthetic Valve Endocarditis
Description: as for outcome 22
Time Frame: 2 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 2.3

45. Other Pre Specified Outcome: Incidence of Prosthetic Valve Thrombosis
Description: as for outcome 25
Time Frame: 2 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0.0

46. Other Pre Specified Outcome: Valve-related Dysfunction
Description: as for outcome 28
Time Frame: 2 Year
Population: Number of implanted subjects with evaluable site-reported echo data
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 23
Participants | 0.0

47. Other Pre Specified Outcome: Incidence of Valve-related Dysfunction Requiring Repeat Procedure
Description: Incidence of Valve-related dysfunction requiring repeat procedure
Time Frame: 2 Year
Population: Number of attempted implant population
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 50
Percent of Participants (K-M Rate) | 0.0

48. Other Pre Specified Outcome: Valve Hemodynamic Performance Metric - Mean Aortic Gradient
Description: Mean aortic gradient
Time Frame: 2 year
Population: Number of implanted subjects with site reported echo evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 25
mmHg | 9.8 (5.0)

49. Other Pre Specified Outcome: Valve Hemodynamic Performance Metric - Effective Orifice Area
Description: Effective orifice area
Time Frame: 2 year
Population: Number of implanted subjects with site reported echo evaluable data
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 23
cm^2 | 1.73 (0.47)

50. Other Pre Specified Outcome: Valve Hemodynamic Performance Metric - Degree of Aortic Regurgitation (Transvalvular, Paravalvular, Total)
Description: Degree of aortic regurgitation (transvalvular, paravalvular, total)
Time Frame: 2 year
Population: Number of implanted subjects with site reported echo evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Total Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System | Paravalvular Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System | Transvalvular Aortic Regurgitation - Experimental: Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 26 | 26 | 26
Participants
  None | 11 | 12 | 21
  Trace | 7 | 7 | 3
  Mild | 8 | 7 | 2
  Mild to Moderate | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Moderate to Severe | 0 | 0 | 0
  Severe | 0 | 0 | 0

51. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Classification
Description: as for outcome 35
Time Frame: 2 Year
Population: Number of attempted subjects with available NYHA
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic CoreValve™ Evolut™ PRO System
Number analyzed (Participants) | 41
Participants
  NYHA I | 7
  NYHA II | 24
  NYHA III | 5
  NYHA IV | 0.0
  Died Prior to visit | 5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected throughout the study duration, starting at the time of written informed consent signed. Adverse event data are currently available and reported for 2 year post-procedure.
Description: All AEs that occur during the study need to be collected by investigator or designee.
Arm/Group | Experimental: Medtronic CoreValve™ Evolut™ PRO System
All-Cause Mortality (participants affected / at risk) | 5/50
Serious Adverse Events (participants affected / at risk) | 28/50
Other Adverse Events (participants affected / at risk) | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Medtronic CoreValve™ Evolut™ PRO System (N=50)
Atrioventricular block complete (Cardiac disorders) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Coronary ostial stenosis (Cardiac disorders) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Blood pressure decreased (Investigations) | 1 (1)
PaO2/FiO2 ratio decreased (Investigations) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 3 (4)
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1)
Cholangitis Infective (Infections and infestations) | 1 (1)
Coronavirus Pneumonia (Infections and infestations) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urethritis (Infections and infestations) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shoulder Fracture (Injury, poisoning and procedural complications) | 2 (2)
Endocarditis Bacterial (Infections and infestations) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 1 (1)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Medtronic CoreValve™ Evolut™ PRO System (N=50)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 6 (6)
Bundle branch block left (Cardiac disorders) | 14 (14)
Myocardial injury (Cardiac disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 60 days of receipt Medtronic (MDT) will verify presence of Confidential Information (CI) & won't censor or interfere with presentation/conclusions except to protect CI (other than Study Data) & its rights in patentable or copyrightable materials, & check technical accuracy of MDT data.

If told by MDT that Publication contains CI or technical errors of MDT data, PI will make requested changes before publishing/presenting. PI will delay publication up to 90 more days, if requested.

DOCUMENTS (6):
  • Study Protocol: Study Protocol V4.0 (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04982588/Prot_000.pdf
  • Study Protocol: Study Protocol V3.0 (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04982588/Prot_001.pdf
  • Study Protocol: Study Protocol V2.0 (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04982588/Prot_002.pdf
  • Study Protocol: Study Protocol V5.0 (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04982588/Prot_004.pdf
  • Statistical Analysis Plan: V2.0 (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04982588/SAP_003.pdf
  • Statistical Analysis Plan: V3.0 (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04982588/SAP_005.pdf